CLINICAL TRIAL: NCT07213206
Title: Chemotherapy Omission in HR-positive/HER2-positive Breast Cancer With Lymph Node Negative Disease Receiving Adjuvant Endocrine Therapy and CDK4/6 Inhibitor Combined With Anti-HER2 Therapy
Brief Title: CDK4/6 Inhibitor Intensification and Chemotherapy De-Escalation for Early-stage Luminal-HER2 Breast Cancer
Acronym: Cinderella
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N095
Record Dates: First submitted 2025-07-18; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDK 4/6 inhibitor combined therapy (omit chemo) (Experimental): CDK4/6 inhibitor for two years combined with endocrine therapy for five years and Trastuzumab(without chemo) for one year
  Interventions: Drug: CDK 4/6 inhibitor combined therapy (omit chemo)
- standard of care (Active Comparator): four cycles of docetaxel and cyclophosphamide or four cycles of weekly paclitaxel combined with Trastuzumab for one year
  Interventions: Drug: standard of care

INTERVENTIONS:
Drug: CDK 4/6 inhibitor combined therapy (omit chemo) — CDK 4/6 inhibitor and endocrine therapy combined with Trastuzumab ( without chemotherapy)
  Arms: CDK 4/6 inhibitor combined therapy (omit chemo)
Drug: standard of care — four cycles of docetaxel and cyclophosphamide or four cycles of weekly paclitaxel Combined with Trastuzumab followed by standard endocrine therapy( aromatase inhibitors or tamoxifen，Ovarian function suppression agents may be added if premenopausal)
  Arms: standard of care

SUMMARY:
The investigators designed a phase III clinical trial involving hormone receptor-positive and HER2-positive stage I breast cancer patients. This trial aims to evaluate the efficacy and safety of a treatment regimen combining CDK4/6 inhibitors, endocrine therapy, and anti-HER2 therapy compared with the traditional approach of chemotherapy combined with anti-HER2 therapy.

DETAILED DESCRIPTION:
For patients with hormone receptor-positive and HER2-positive breast cancer, the NCCN guidelines recommend that those with tumors larger than 1 cm or positive lymph nodes should receive standard adjuvant therapy comprising chemotherapy combined with targeted and endocrine therapy. In contrast, for patients with tumors smaller than 1 cm and negative lymph nodes, endocrine therapy alone or in combination with targeted therapy and chemotherapy may be considered. Therefore, in patients with stage I hormone receptor-positive and HER2-positive breast cancer, it remains unclear whether chemotherapy can be omitted by intensifying endocrine therapy through the addition of CDK4/6 inhibitors, particularly considering the intrinsic therapeutic efficacy of endocrine agents and their potential synergistic interaction with anti-HER2 therapy. To further minimize treatment-related toxicity and identify the optimal adjuvant treatment strategy for patients with HER2-positive stage I breast cancer, the investigators designed a phase III clinical trial involving hormone receptor-positive and HER2-positive stage I breast cancer patients. This trial aims to evaluate the efficacy and safety of a treatment regimen combining CDK4/6 inhibitors, endocrine therapy, and anti-HER2 therapy compared with the traditional approach of chemotherapy combined with anti-HER2 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged between 18 and 75 years;
2. Unilateral invasive carcinoma confirmed by histopathological examination;
3. Postoperative pathological stage I early breast cancer: histologically confirmed invasive carcinoma with a maximum tumor diameter not exceeding 2 cm and no lymph node metastasis (N0);
4. Estrogen receptor (ER) expression ≥ 50%;
5. Immunohistochemical and molecular pathology must meet one of the following criteria: HER-2 overexpression (3+) or HER-2 (0-2+) with gene amplification confirmed by fluorescence in situ hybridization (FISH);
6. Histological grade 1-2 or selected grade 3 tumors with at least one of the following additional features: PAM50 or HER2-based subtyping indicating luminal phenotype , or tumor size ≤ 1 cm );
7. Adequate major organ function, defined as:

(1) Hematologic parameters: hemoglobin (HB) ≥ 90 g/L (without blood transfusion within 14 days), absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L, platelet count (PLT) ≥ 100 × 10⁹/L; (2) Biochemical parameters: total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN, serum creatinine (Cr) ≤ 1 × ULN, and calculated creatinine clearance > 50 mL/min using the Cockcroft-Gault formula; 8) Cardiac function preserved with left ventricular ejection fraction (LVEF) > 50%; 9) Willing to participate in the study, with signed informed consent, good compliance, and willingness to comply with follow-up requirements.

Exclusion Criteria:

1. Tumors with a maximum diameter exceeding 2 cm and/or presence of positive axillary lymph nodes;
2. HER2-negative status defined as HER2- or HER2+ by immunohistochemistry; or HER2 2+ by immunohistochemistry without gene amplification confirmed by fluorescence in situ hybridization (FISH);
3. Patients who have previously received neoadjuvant therapy or any form of systemic or non-surgical local treatment prior to enrollment, including chemotherapy, targeted therapy, radiotherapy, or endocrine therapy;
4. History of other malignant tumors, excluding cured basal cell carcinoma of the skin and cervical carcinoma in situ;
5. Has metastatic (Stage 4) breast cancer;
6. Pregnant or lactating women, as well as women of childbearing potential who are unable to use effective contraception;
7. Patients currently enrolled in other clinical trials;
8. Severe organ dysfunction involving the cardiovascular, pulmonary, hepatic, or renal systems, including left ventricular ejection fraction (LVEF) < 50% as assessed by echocardiography; history of severe cardiovascular or cerebrovascular events within 6 months prior to enrollment (e.g., unstable angina, chronic heart failure, uncontrolled hypertension > 150/90 mmHg, myocardial infarction, or stroke); patients with poorly controlled diabetes mellitus; patients with severe or uncontrolled hypertension;
9. Active severe or uncontrolled infections;
10. Patients with a history of substance abuse involving psychotropic drugs with ongoing dependency, or a documented history of psychiatric disorders that may interfere with study compliance;
11. Patients deemed unsuitable for participation by the principal investigator or designated study physician.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-10-07 (Estimated); Primary Completion 2032-09-01 (Estimated); Study Completion 2035-09-01 (Estimated)

PRIMARY OUTCOMES:
iDFS | 3 years
  invasive disease-free survival

SECONDARY OUTCOMES:
RFS | 3 years
  recurrence-free survival
DRFS | 3 years
  distant recurrence-free survival
OS | 3 years
  overall survival
adverse effects | 3 years
  adverse effects according to CTCAE 5.0